CLINICAL TRIAL: NCT04761549
Title: Identification of Key Parameters to Initiate the Shift Towards 3D, Dynamic and Mechanically-informed Decision Making in Adolescent Idiopathic Scoliosis
Brief Title: 3D, Dynamic and Mechanically-informed Decision Making in AIS
Acronym: 3D-AIS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S64400
Record Dates: First submitted 2021-02-15; First posted 2021-02-21 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-06

CONDITIONS: Adolescent Idiopathic Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adolescent Idiopathic Scoliosis (Other): Questionnaires, Radiological EOS scan, 3D Dynamic Motion analysis
  Interventions: Procedure: Adolescent Idiopathic Scoliosis

INTERVENTIONS:
Procedure: Adolescent Idiopathic Scoliosis — Adolescent Idiopathic Scoliosis

SUMMARY:
Adolescent Idiopathic Scoliosis (AIS) is a growth defect of the spine that primarily occurs in prepubertal children between the age of 10 to 14 years, affecting approximately 3% of these otherwise normal children. AIS has been associated with problems related to posture, load-related back pain, as well as aesthetic problems, e.g. the induced asymmetry of the shoulder. Therefore, early diagnosis followed by the appropriate treatment is vital to prevent further curve progression of AIS and minimize the health-related complications of these patients.

The current treatment recommendation to stop curve progression for an immature patient with a scoliosis curve between 25 and 40 degrees is to wear a brace. If the curve in the skeletally immature patient is not responding to the brace treatment, dynamic scoliosis correction by vertebral body tethering can be considered when there is still some growth potential left. State-of-the-art guidelines for the selection of fusion levels are currently mainly based on two-dimensional (2D) static radiographic parameters (such as, the Cobb angle and Shoulder balance) and a qualitative assessment of 2D bending or traction radiographs. Several classification systems and algorithms that are based on the 2D static radiographic (X-ray) parameters exist to assist surgeons in determining the appropriate levels to be instrumented. Despite this wide range of classification systems and detailed guidelines available in the literature, spinal fusion does not always yield satisfying 2D radiographic clinical outcome, with revision rates ranging from 3.9% to 22%.

Overall, the surgeon is presently not provided with 3D dynamic and mechanical information regarding the deformity of the AIS to guide the decision-making. Obtaining this vital 3D dynamic information regarding the curvature and mechanical behavior of the spine will allow the surgeon to make an evidence-based and well-informed decisions in the treatment of the AIS patient. Consequently, realizing these objectives has the potential to improve patient satisfaction, reduce the postoperative complications and accordingly reduce socio-economic costs associated with AIS treatment. Recent advances in the use of subject specific musculoskeletal models will form the basis to realize this shift from 2D to 3D dynamic in AIS care.

DETAILED DESCRIPTION:
Adolescent Idiopathic Scoliosis (AIS) is a growth defect of the spine that primarily occurs in prepubertal children between the age of 10 to 14 years, affecting approximately 3% of these otherwise normal children. The spine, which is normally straight in a posterior view, forms one or two lateral curves with associated turns around its longitudinal axis, like a spiral staircase. AIS has been associated with problems related to posture, load-related back pain, as well as aesthetic problems, e.g. the induced asymmetry of the shoulder. Therefore, early diagnosis followed by the appropriate treatment is vital to prevent further curve progression of AIS and minimize the health-related complications of these patients.

The current treatment recommendation to stop curve progression for an immature patient with a scoliosis curve between 25 and 40 degrees is to wear a brace. If the curve in the skeletally immature patient is not responding to the brace treatment, dynamic scoliosis correction by vertebral body tethering can be considered when there is still some growth potential left. This recent (2019) US Food and Drug Administration (FDA) approved device for tethering gradually corrects the scoliosis by slowing growth on the convex side of the curve. This technique is minimally invasive, preserves motion, and does not preclude spinal fusion surgery when unsuccessful, but at the moment long term results are lacking. When a curve reaches 50 degrees, it's clinically expected to further progress and further growth potential is low, a "scoliosis fusion" surgery is recommended. This type of surgery permanently attaches all vertebrae in the area to be corrected to each other by surgical instrumentation. In order to reach the desired surgical outcome, one of the main decisions to be made by the treating surgeon is the selection of the appropriate fusion levels (i.e. the upper and lower instrumented vertebra). State-of-the-art guidelines for the selection of fusion levels are currently mainly based on two-dimensional (2D) static radiographic parameters (such as, the Cobb angle and Shoulder balance) and a qualitative assessment of 2D bending or traction radiographs. Several classification systems and algorithms that are based on the 2D static radiographic (X-ray) parameters exist to assist surgeons in determining the appropriate levels to be instrumented. Despite this wide range of classification systems and detailed guidelines available in the literature, spinal fusion does not always yield satisfying 2D radiographic clinical outcome, with revision rates ranging from 3.9% to 22%. Besides an adequate correction of the spinal curve in all three planes, factors such as shoulder level, clinical rib and lumbar hump, as well as scar size, play a major role in the evaluation of treatment success. This contributes to the fact that spinal fusion in AIS patients is a costly procedure. Therefore, the potential limitations of the current state-of-the-art surgical decision making should be critically examined and improved where possible.

There are three main limitations of the state-of-the-art classification systems highlighted in the literature. The first limitation is that classification systems use 2D static radiographic parameters to provide guidelines for a three-dimensional (3D) deformity of the spine. The second limiting factor is that the current classification systems do not include dynamic components. Even though, it has been shown that a 2D radiographic assessment is not representative of spinal balance during daily life activities. The third limitation is that the surgeon has only limited information on the mechanical behavior of the patient's spine. Mechanical information of the spine, such as the spine stiffness (i.e. a measure of the force required to deform a patient's spine), is critical for the selection of the appropriate fusion levels that, for example, would result in balanced shoulders.

Overall, the above highlighted limitations indicate that the surgeon is presently not provided with 3D dynamic and mechanical information regarding the deformity of the AIS to guide the decision-making. Consequently, there is an immediate need to overcome this apparent gap in the decision-making in AIS by identifying the key parameters that provide the surgeon with vital 3D dynamic information regarding the deformity. Obtaining this vital 3D dynamic information regarding the curvature and mechanical behavior of the spine will allow the surgeon to make an evidence-based and well-informed decisions in the treatment of the AIS patient. Consequently, realizing these objectives has the potential to improve patient satisfaction, reduce the postoperative complications and accordingly reduce socio-economic costs associated with AIS treatment. Recent advances in the use of subject specific musculoskeletal models will form the basis to realize this shift from 2D to 3D dynamic in AIS care.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with Adolescent Idiopathic Scoliosis
* 10-35 years old
* Patient is scheduled to be surgically treated by vertebral body tethering (VBT) or selective fusion at UZ Leuven
* Informed consent obtained: also from parent/guardian in case of minors

Exclusion Criteria:

* Patient has undergone a fusion or VBT procedure before
* Patient has a severe underlying illness which might influence the outcome of the surgery
* Making it reasonable for the investigator to exclude the patient

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-19 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
3D dynamic parameters | up to 2 years post-operatively
  The key 3D dynamic parameters that have the potential to improve the clinical decision-making in AIS specifically with regards to shoulder balance and PROMs will be identified from the wide range of data collected at the different timepoints of the present study. The specific parameters to be included in the analysis will be partially informed by the 3D parameters identified from our ongoing retrospective study.

SECONDARY OUTCOMES:
Biomechanically-informed Adolescent Idiopathic Scoliosis specific 3D model | up to 2 years post-operatively
  The development of a biomechanically-informed AIS specific 3D model will allow us to calculate the parameters of interest at different timepoints. This information could additionally be used to investigate the compensations made by the AIS patients after surgery during static and dynamic activities. Furthermore, the developed 3D model could in the future be used to examine the possibility of integrating computational simulations at different timepoints in the treatment (e.g. pre- and preoperative), which are a safe non-invasive method to gain knowledge about the consequences of the surgery on the patient in a virtual environment.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastiaan Schelfaut, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No